CLINICAL TRIAL: NCT04453761
Title: Thiamine Influenced on Substrate Energy Effectiveness in Indonesian Children Undergoing Congenital Heart Disease Surgery With Cardiopulmonary Bypass Procedure and Oral Thyroid Supplementation
Brief Title: Thiamine Influenced on Substrate Energy Effectiveness in Indonesian Children Undergoing Cardiopulmonary Bypass
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Cardiovascular Center Harapan Kita Hospital Indonesia (Other)
Responsible Party: Principal Investigator, Eva M Marwali,MD, Eva M Marwali, MD, Phd, National Cardiovascular Center Harapan Kita Hospital Indonesia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LB.02.01/VII/225/KEP.066/2017
Record Dates: First submitted 2018-04-10; First posted 2020-07-01 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: Thiamine Deficiency; Congenital Heart Disease; Cardiopulmonary Bypass
Keywords: thiamine supplementation; congenital heart disease; paediatric cardiac surgery; cardiopulmonary bypass
MeSH Terms: conditions — Thiamine Deficiency; Heart Defects, Congenital | interventions — Vitamin B Complex; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drugs Group (Experimental): Thiamine IV
  Interventions: Drug: Neurobion
- Placebo (Placebo Comparator): NaCl IV
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Neurobion — Intravenous Thiamine 2 mg/kg in Neurobion injection
  Other Names: Vitamin B1 IV
  Arms: Drugs Group
Drug: Placebo — Intravenous NaCl0.9%
  Other Names: NaCl 0.9%
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, controlled trial design. It was conducted with a main purpose of evaluating the effect of thiamine supplementation on serum lactate and lactate-pyruvate ratio after surgery as direct indicators of tissue perfusion and indirect markers of energy substrate availability for effective mitochondrial function and intubation time as clinical outcome.

DETAILED DESCRIPTION:
All patients who undergo open cardiac surgery for their congenital heart disease on the research period will be recruited consecutively and evaluated according to the study criteria. Parents or guardians were explained about the procedure. Agreement will be concluded by signing the informed consent. Baseline data including age, nutritional status, diagnosis, types of heart disease (cyanotic or acyanotic), restrictive or non restrictive pulmonary blood flow heart disease, pre-surgical peripheral saturation, pulmonary hypertension and any syndromes associated with heart disease will be recorded on the study sheets.

Patients will be randomised using block randomisation procedure with a block size of 4 on treatment and control group. Included participants will be marked by specific randomisation number by a research assistant physician who is not involved in patients' management. A pharmacist will acquire and open a prepared envelope containing the randomisation number. The patients, parents/guardians, research physicians, other physicians or paramedics involved in patients' treatment will be blinded.

Placebo (Intravenous Normal Saline) and intravenous thiamine (2 mg/kg) will be administered at induction time, 1 hours after surgery and once everyday for three days by pharmacist according to randomization result. All subject are given oral T3 supplementation (1 mcg/kg) every 6 hours by pharmacist as research protocol. Oral T3 supplementations are given every 6 hours, started from induction time until 11 doses (60 hours until the first dose). Drugs is diluted with 2.5 cc aqua and administerednisterd using nasogastric tube.

Blood will be withdrawn from arterial line access for 2.5 cc in order to test thiamine, lactate, and pyruvate concentration, as well as, measuring LDH and PDH activity. Thiamine will be examined from blood plasma using liquid chromatography tandem mass spectometry. Thiamine concentration below ≤ 7 nmol/L is considered low. PDH will be examined from Peripheral Blood Mononuclear Cells (PBMCs) which will be isolated from fresh blood. PDH activity will be tested after breaking cell membrane to initiate mitochondria lysis, this process will be done by immunocapture and micro-plate based assay. Lactate and pyruvate measurement will be tested using an enzymatic kit specific for lactate and pyruvate called Sigma Aldrich reagent. Thiamine concentration, lactate concentration, pyruvate concentration, LDH and PDH activity is going to be measured at 4 time; induction time, one hour, 24 hours, 72 hours after aortic clamp removal.

Measurement of blood gas analysis, blood glucose, central vein saturation and oxygen extraction ratio will be performed at induction time, 1 hours, and 12 hours post-surgery.

Organ functions evaluation was performed by serially measuring SGOT and SGPT (liver function) as well as ureum and creatinine (renal function) on ICU admission.

Echocardiography evaluation will be done on the first, second and third day after surgery to assess the patient's ejection fraction, stroke volume, cardiac volume and index, tricuspid annular plane systolic excursion (TAPSE), left heart diastolic functions and SVRI calculation. It will be done by 2 research cardiologists.

Post-surgical managements will be decided according to the paediatric ICU National Cardiovascular Center Harapan Kita treatment protocols. Inotropic concentration will be evaluated by inotropic and vasoactive-inotropic scoring every 6 hours in the first 24 hours and every 12 hours after the second and third 24 hours. The amount of diuretics used will be calculated 72 hours after ICU admission. Peritoneal dialysis and continuous veno-venous hemofiltration (CVVH) is going to be assessed by means of the length of therapy, renal function and fluid balance. Decision to extubate will be carried out by a physician responsible according to the treatment protocols. Every reintubation is going to be recorded as number and length of intubation. The length of ICU and hospital stay and mortality will be evaluated in both study groups.

Operative data such as Aristotle score, residual lesions presence, open thorax on ICU admission, CPB duration, Aox duration and a number of procedures during CPB including ultrafiltration, hypothermia and hemodilution is going to be recorded in the research sheets. History of medication used which may interfere with the function of thyroid such as steroids, dopamine and amiodarone will also be recorded.

There will be one physician who know the subject's allocation. This physician is not involve in any kind of patients' treatment and act as the study supervisor to evaluate if any suspicion on drug adverse reactions occurred. Drug adverse reaction is going to be monitored by evaluating heart rhythm, heart rate, blood pressure and peripheral temperature for every 6 hours in the first 24 hours and every 12 hours in the second and third 24 hours of ICU treatment. The criteria of drug adverse reaction are stated in the adverse effects form; they are tachycardia, arrhythmia, hypertension and refractory hyperthermia. Any suspicion of the presence of drug adverse effect is going to be recorded in the form and reported to the supervising doctor for further analysis. Management on this reaction will be done by the ICU treating doctor

ELIGIBILITY:
Inclusion Criteria:

All patients with congenital heart disease, 2 years old or less, with moderate to severe malnutrition are included. Types of congenital heart disease suffered required subject to undergo surgery using cardiopulmonary bypass machine with Aristotle score of 6-9.

Exclusion Criteria:

1. Body weight of less than 2 kg at the study period
2. Suffering from pre-surgical tachyarrhythmia or other types of arrhythmias
3. Pre-surgical sepsis
4. Serum creatinine of more than 2 mg/dL
5. Diagnosed with thyroid abnormalities prior to the surgery

Ages: 1 Month to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate the effect of thiamine supplementation to pyruvate levels | at 6 hours post cross clamp removal
  Comparing the lab parameter indicate pyruvate levels

SECONDARY OUTCOMES:
Evaluate the effect of thiamine supplementation to cardiac output. | Within 1 days of surgery
  Measuring Cardiac output

CONTACTS AND LOCATIONS:
Overall Officials: Eva M Marwali, MD, PhD, Principal Investigator — National Cardiovascular Centre Harapan Kita Jakarta Indonesia
Locations (1):
- National Cardiovascular Center Harapan Kita, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Marwali EM, Boom CE, Budiwardhana N, Fakhri D, Roebiono PS, Santoso A, Sastroasmoro S, Slee A, Portman MA. Oral Triiodothyronine for Infants and Children Undergoing Cardiopulmonary Bypass. Ann Thorac Surg. 2017 Aug;104(2):688-695. doi: 10.1016/j.athoracsur.2017.01.001. Epub 2017 Feb 6. PMID 28185643
- [Result] Marwali EM, Boom CE, Sakidjan I, Santoso A, Fakhri D, Kartini A, Kekalih A, Schwartz SM, Haas NA. Oral triiodothyronine normalizes triiodothyronine levels after surgery for pediatric congenital heart disease*. Pediatr Crit Care Med. 2013 Sep;14(7):701-8. doi: 10.1097/PCC.0b013e3182917f87. PMID 23842591
- [Result] Luger M, Hiesmayr M, Koppel P, Sima B, Ranz I, Weiss C, Konig J, Luger E, Kruschitz R, Ludvik B, Schindler K. Influence of intravenous thiamine supplementation on blood lactate concentration prior to cardiac surgery: A double-blinded, randomised controlled pilot study. Eur J Anaesthesiol. 2015 Aug;32(8):543-8. doi: 10.1097/EJA.0000000000000205. PMID 26066773